CLINICAL TRIAL: NCT02276261
Title: The Effect of Vertical Versus Horizontal Vaginal Cuff Closure on Vaginal Length After Laparoscopic Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bridgeport Hospital (Other)
Responsible Party: Principal Investigator, Amanda Tower, Fellow, Bridgeport Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 111401
Record Dates: First submitted 2014-10-20; First posted 2014-10-28 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Hysterectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vertical (Experimental): Vaginal cuff closure performed in a vertical manner.
  Interventions: Procedure: Vaginal cuff closure - vertical
- Horizontal (Active Comparator): Vaginal cuff closure performed in a horizontal manner.
  Interventions: Procedure: Vaginal cuff closure - horizontal

INTERVENTIONS:
Procedure: Vaginal cuff closure - vertical — Vaginal cuff is closed vertically.
  Arms: Vertical
Procedure: Vaginal cuff closure - horizontal — Vaginal cuff is closed horizontally.
  Arms: Horizontal

SUMMARY:
This study has been designed as a prospective randomized trial to be performed at Bridgeport Hospital. Patients planning to undergo a laparoscopic or robotically assisted total laparoscopic hysterectomy with or without removal of adnexal structures will be recruited by the Bridgeport Hospital Minimally Invasive Gynecologic Surgery fellows during their preoperative office visit at the Bridgeport Hospital Gynecologic Oncology office. If enrolled, they will be assigned a sequential study identification number. During their preoperative exam, a baseline POP-Q will be performed. Demographic information will be recorded from the electronic medical record.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing laparoscopic or robotic-assisted laparoscopic hysterectomy
* Under the care of Dr. Dan-Arin Silasi or Dr. Masoud Azodi at Bridgeport Hospital
* Planning to follow up at the Gynecologic Oncology office at Bridgeport Hospital
* Age 18 or older
* Able to give informed consent to participate in the research study

Exclusion Criteria:

* Age less than 18
* Unable to give informed consent
* Patients undergoing radical hysterectomy
* Patients receiving vaginal cuff radiation within the study period
* Patients undergoing concomitant pelvic floor or vaginal suspension procedure

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2014-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Vaginal length | 1-3 weeks postop
  Vaginal length will be measured in cm by standard POP-Q measurements

SECONDARY OUTCOMES:
Vaginal length | 3-4 months postop
  Vaginal length will be measured in cm by standard POP-Q measurements
Cuff closure time | intra-op
  Time will be recorded by the circulating nurse in seconds

OTHER OUTCOMES:
Complications | Up to 4 months post-op
  Including urinary retention, bladder injury, ureteral injury, cuff dehiscence, cuff bleeding requiring further procedures or cauterization

CONTACTS AND LOCATIONS:
Locations (1):
- Bridgeport Hospital, Bridgeport, Connecticut, United States